CLINICAL TRIAL: NCT06911905
Title: Efficacy of Nutritional Supplements on Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fei Li (Other)
Responsible Party: Sponsor-Investigator, Fei Li, Chief Physician, Doctoral Supervisor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHEC-C-2024-086-2
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Dietary Supplements; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional supplements plus treatment as usual (TAU) (Experimental): Participants in experimental group with received nutritional supplements, along with treatments as usual (i.e. behavioral interventions)
  Interventions: Dietary Supplement: Nutritional supplements; Behavioral: Treatment as usual (TAU)
- Treatment as usual (TAU) (Other): Participants in the control group will undergo treatments as usual, such as behavioral interventions
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Dietary Supplement: Nutritional supplements — The nutritional supplements, including Vitamin B1, Vitamin B2, folic acid, Mecobalamin, Vitamin D3, Choline, and Coenzyme Q10, will be administered for a period of three months.
  Arms: Nutritional supplements plus treatment as usual (TAU)
Behavioral: Treatment as usual (TAU) — Participants will undergo treatment as usual, such as behavioral interventions

SUMMARY:
The goal of this clinical trial is to learn if nutritional supplements could alleviate the clinical symptoms in children with autism spectrum disorder. It will also learn about the safety of these nutritional supplements.

Researchers will compare the combination of nutritional supplements and behavioral intervention, to behavioral intervention alone, to see if nutritional supplements work to treat autism.

Participants will receive the combination of nutritional supplements and behavioral interventions or solely behavioral interventions for 3 months. And they will visit the clinic at the beginning of the trial (baseline) and after the 3-month intervention period for examinations.

DETAILED DESCRIPTION:
This is an open-label clinical trial aimed at investigating whether nutritional supplements could alleviate the clinical symptoms in children with autism spectrum disorder. Participants will be randomly assigned to either the experimental group or the control group.

Participants in the experimental group will receive the combination of nutritional supplements, including Vitamin B1, Vitamin B2, folic acid, Mecobalamin, Vitamin D3, Choline, and Coenzyme Q10, along with the behavioral interventions, for a period of three months. Participants in the control group will only undergo behavioral interventions.

during the intervention period, the clinical symptoms, metabolomics of bio-specimens, and potential adverse effects will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2.5 and 6 years old
* Meeting the ASD diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Meeting the ASD diagnostic criteria of the Diagnostic Observational Scale for Autism, Second Edition (ADOS-2）
* CARS total score ≥ 30
* Obtaining informed consent from the legal guardian

Exclusion Criteria:

* History of neurological diseases such as epilepsy
* History of congenital diseases such as hearing, visual impairment
* Diagnosed with metabolic disorders such as hypophosphatemic rickets
* Diagnosed with genetic or chromosomal abnormalities
* Brain structural abnormalities detected by MRI which required surgical intervention
* Currently participating in other clinical trials
* Received any new intervention within 8 weeks prior to enrollment

Ages: 30 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, Second Edition (SRS-2) | From enrollment to the end of treatment at 3 months
  Social Responsiveness Scale, Second Edition (SRS-2) is a scale used to evaluate the presence and severity of social impairment. The scores of the SRS-2 rate from 0 to 195, and higher scores indicate more severe symptoms. Changes of the SRS-2 scores from baseline to 3 month after treatment will be analyzed to assess the effect of the intervention on children with autism spectrum disorder.

SECONDARY OUTCOMES:
Clinical Global Impressions Scale (CGI) | From enrollment to the end of treatment at 3 months
  Clinical Global Impressions Scale (CGI) is a scale used to assess the severity of the illness and the global improvement of the participants under intervention.The Clinical Global Impression - Severity scale (CGI-S) is a clinician rated 7-point measure of overall severity. Scores range from 1 (Normal, not at all ill) through 4 (Moderately ill) to 7 (Among the most extremely ill patients). The Clinical Global Impression - Improvement scale (CGI-I) is the companion measure that evaluates the change in the patient's symptoms relative to baseline. Scores range from 1 (Very much improved) through 4 (No Change) to 7 (Very much worse).
Childhood Autism Rating Scale (CARS) | From enrollment to the end of treatment at 3 months
  CARS is a behavior-rating scale used to assess the presence and severity of the symptoms associated autism spectrum disorder. The scores of the CARS rate from 15 to 60, and higher scores indicate more severe symptoms. The changes in the CARS scores from baseline to 3 months after the treatment will be analyzed to assess the impact of the intervention on participants with autism spectrum disorder
Aberrant Behavior Checklist (ABC) | From enrollment to the end of treatment at 3 months
  Aberrant Behavior Checklist (ABC) is a 58-item instrument used to measure behavior problems across five sub-scales: hyperactivity, irritability, social withdrawal, stereotypic behavior and inappropriate speech. Each item rates behavior severity on a 4 point scale from 0 (Not at all a problem) to 3 (The problem is severe in degree). A higher score indicates more frequent aberrant behaviors.Changes of the total scores and scores of subscales from baseline to 3 month after treatment will be analyzed.
Chinese Communicative Development Inventory (CCDI) | From enrollment to the end of treatment at 3 months
  Chinese Communicative Development Inventory (CCDI) is a questionnaire used to measures the language abilities. Higher scores suggest better language level. The changes in the CCDI between baseline and 3 month after treatment will be analyzed.

OTHER OUTCOMES:
Metabolomics tests | From enrollment to the end of treatment at 3 months
  Biological specimens such as blood, urine, and faecal samples will be collected at baseline and at the 3-month follow-up. These samples will be used for metabolomic testing and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, MD, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The Study Protocol, Statistical Analysis Plan, Informed Consent Form, and other relevant documents will be available under reasonable and ethically approved request to the corresponding authors.